CLINICAL TRIAL: NCT02528942
Title: Early Phase Clinical Trial Incorporating Lung Function Imaging Into Radiation Therapy for Lung Cancer Patients
Brief Title: Feasibility Study Incorporating Lung Function Imaging Into Radiation Therapy for Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-1856.cc; 1R01CA200817-01 (NIH)
Record Dates: First submitted 2015-08-06; First posted 2015-08-19 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Lung Neoplasms; Lung Cancer
Keywords: Lung cancer; Radiation therapy; 4DCT-ventilation imaging
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation therapy (Experimental): The functional avoidance radiation therapy plan will be delivered using a standard course of radiation treatment on a linear accelerator. Patients will receive daily radiation treatment for 15-35 days.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy will be given to study patients.

SUMMARY:
The proposed study is in the field of thoracic radiation oncology where radiation therapy is used to treat lung cancer. The primary objective of the early phase clinical trial will be to evaluate the safety of performing functional avoidance radiation therapy for lung cancer patients using 4D computed tomography (4DCT) ventilation imaging.

DETAILED DESCRIPTION:
This study plans to learn more about radiation therapy. Radiation therapy is one of the main treatments used to treat lung cancer. One of the known side effects of this radiation therapy is scarring of the lungs and reduced lung function that can result in shortness of breath. At this time the radiation treatment plan does not take into account differences in lung function between one part of the lung and another. Studies have shown that lung function can vary substantially throughout the lungs. This study aims to plan the radiation therapy to be away from the highest functioning portions of lungs while still delivering the intended radiation dose to the tumor. This study will allow researchers to determine whether taking lung function information into account when designing radiation treatment plans can protect lung function after radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of pathologically confirmed lung cancer by tumor biopsy and/or fine-need aspiration
2. Lung Cancer patients that will undergo definitive radiation therapy defined as 45-75 Gy as part of standard of care for their disease
3. 18 years of age or older
4. Signed informed consent
5. Planned curative intent chemotherapy, delivered concurrently or sequentially in combination with radiotherapy
6. The patient's 4DCT-ventilation image meets image heterogeneity criteria

Exclusion Criteria:

1. Patients receiving Stereotactic Body Radiation Therapy
2. Patient receiving palliative radiation therapy (defined as less than 45 Gy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yevgeniy Vinogradskiy, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Beaumont Health System, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poiset SJ, Lombardo J, Castillo E, Castillo R, Jones B, Miften M, Kavanagh B, Dicker AP, Boyle C, Simone NL, Movsas B, Grills I, Rusthoven CG, Vinogradskiy Y, Wilson L. Patient-Reported Outcomes: Comparing Functional Avoidance and Standard Thoracic Radiation Therapy in Lung Cancer. JCO Clin Cancer Inform. 2025 Feb;9:e2400202. doi: 10.1200/CCI-24-00202. Epub 2025 Feb 4. PMID 39903899
- [Derived] Porter EM, Myziuk NK, Quinn TJ, Lozano D, Peterson AB, Quach DM, Siddiqui ZA, Guerrero TM. Synthetic pulmonary perfusion images from 4DCT for functional avoidance using deep learning. Phys Med Biol. 2021 Aug 23;66(17). doi: 10.1088/1361-6560/ac16ec. PMID 34293726

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy
Started | 101
Completed | 67
Not Completed | 34
Not completed — Did not meet imaging criteria | 9
Not completed — Lost to Follow-up | 25

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 67
Age, Continuous [Median (Full Range); unit: years] | 66 [44 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 64
  More than one race | 0
  Unknown or Not Reported | 0
Karnofsky Performance Scale (KPS) [Median (Full Range); unit: units on a scale] — The Karnofsky Performance Scale (KPS) is a common performance status assessment tool in Oncology for predicting of length of survival in terminally ill patients. The KPS is an 11 point rating scale which ranges from normal functioning (100) to dead (0) in ten point increments. Use of these 11 points is necessary, meaning that estimates between points cannot be made.
  units on a scale | 90 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Radiation Safety (Rate of Grade 2 or Higher (Grade 2+) Radiation Pneumonitis as Defined by the Common Toxicity Criteria for Adverse Effects (CTCAE) Scoring System
Description: To assess safety, investigators will evaluate the rate of grade 2 or higher (grade 2+) radiation pneumonitis as defined by the Common Toxicity Criteria for Adverse Effects (CTCAE) scoring system.
Time Frame: Up to 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 67
Participants | 10

2. Secondary Outcome: Percentage of Patients Eligible for 4DCT-ventilation Functional Avoidance
Description: The percentage will be calculated by taking the ratio of patients that had lung function profiles suitable for functional avoidance and patients that were clinically eligible (receiving 45-75 Gy).
Time Frame: Up to 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 67
Participants | 9

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 12/67
Serious Adverse Events (participants affected / at risk) | 10/67
Other Adverse Events (participants affected / at risk) | 8/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (N=67)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Espophagitis (Gastrointestinal disorders) | 2 (2)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
fever (Infections and infestations) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
near syncope (Nervous system disorders) | 1 (1)
Weight loss (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (N=67)
Esophagitis (Gastrointestinal disorders) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT02528942/Prot_SAP_000.pdf